CLINICAL TRIAL: NCT01250418
Title: A Comparison Between the Correlation of the Bispectral Index Versus Snap Index With the Observer's Assessment of Alertness and Sedation (OAA/S) Scale During a Sedation Regimen With and Without Ketamine
Brief Title: SNAP VS BIS(OAA/S) Scale During a Sedation Regimen With and Without Ketamine
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Monitor manufacturer stopped marketing plan for the product.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Gildasio De Oliveira, Gildasio De Oliveira, M.D. Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: STU00031783
Record Dates: First submitted 2010-08-03; First posted 2010-11-30 (Estimated); Results first posted 2014-08-28 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Pain
Keywords: Bispectral Index; Ketamine
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine Group (Active Comparator): ketamine bolus of 0.25mg/kg followed by an infusion set at 1.5 mcg /kg/min.
  Interventions: Drug: Ketamine group
- No ketamine (No Intervention): No ketamine added to anesthesia regimen

INTERVENTIONS:
Drug: Ketamine group — ketamine bolus of 0.25mg/kg followed by an infusion set at 1.5 mcg /kg/min.
  Arms: Ketamine Group

SUMMARY:
The study question: Does the SNAP-Index (SI) correlates better with the OASS than the BIS Monitor during sedation with ketamine?

The study hypothesis: Since the SNAP II monitor seems to be more responsive during emergence of anesthesia, it will have a better correlation with the OASS than the BIS monitor with the use of ketamine.

ELIGIBILITY:
Inclusion Criteria:

* Age : 18-64 years
* ASA : I-III
* Procedure : Breast or gynecological surgery
* Anesthesia :Monitored anesthesia care

Exclusion Criteria:

* Pregnancy
* Breast Feeding
* Body Mass Index >35kg/m2
* Drug or Alcohol abuse
* Use anticonvulsants
* History of CVA
* Drop-out criteria:

  * Patient or surgeon request
  * Conversion to general anesthesia
  * Inability to obtain data from both monitors

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2010-08; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gildasio DeOliveira, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

REFERENCES:
- [Background] Chernik DA, Gillings D, Laine H, Hendler J, Silver JM, Davidson AB, Schwam EM, Siegel JL. Validity and reliability of the Observer's Assessment of Alertness/Sedation Scale: study with intravenous midazolam. J Clin Psychopharmacol. 1990 Aug;10(4):244-51. PMID 2286697
- [Background] Sigl JC, Chamoun NG. An introduction to bispectral analysis for the electroencephalogram. J Clin Monit. 1994 Nov;10(6):392-404. doi: 10.1007/BF01618421. PMID 7836975
- [Background] Glass PS, Bloom M, Kearse L, Rosow C, Sebel P, Manberg P. Bispectral analysis measures sedation and memory effects of propofol, midazolam, isoflurane, and alfentanil in healthy volunteers. Anesthesiology. 1997 Apr;86(4):836-47. doi: 10.1097/00000542-199704000-00014. PMID 9105228
- [Background] Iselin-Chaves IA, Flaishon R, Sebel PS, Howell S, Gan TJ, Sigl J, Ginsberg B, Glass PS. The effect of the interaction of propofol and alfentanil on recall, loss of consciousness, and the Bispectral Index. Anesth Analg. 1998 Oct;87(4):949-55. doi: 10.1097/00000539-199810000-00038. PMID 9768800
- [Background] Song D, Joshi GP, White PF. Titration of volatile anesthetics using bispectral index facilitates recovery after ambulatory anesthesia. Anesthesiology. 1997 Oct;87(4):842-8. doi: 10.1097/00000542-199710000-00018. PMID 9357886
- [Background] Sebel PS, Lang E, Rampil IJ, White PF, Cork R, Jopling M, Smith NT, Glass PS, Manberg P. A multicenter study of bispectral electroencephalogram analysis for monitoring anesthetic effect. Anesth Analg. 1997 Apr;84(4):891-9. doi: 10.1097/00000539-199704000-00035. PMID 9085977
- [Background] Dressler O, Schneider G, Stockmanns G, Kochs EF. Awareness and the EEG power spectrum: analysis of frequencies. Br J Anaesth. 2004 Dec;93(6):806-9. doi: 10.1093/bja/aeh270. Epub 2004 Sep 17. PMID 15377585
- [Background] Wong CA, Fragen RJ, Fitzgerald P, McCarthy RJ. A comparison of the SNAP II and BIS XP indices during sevoflurane and nitrous oxide anaesthesia at 1 and 1.5 MAC and at awakening. Br J Anaesth. 2006 Aug;97(2):181-6. doi: 10.1093/bja/ael131. Epub 2006 May 23. PMID 16720676

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketamine Group | No Ketamine
Started | 9 | 16
Completed | 8 | 15
Not Completed | 1 | 1
Not completed — monitor data failure | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine Group | No Ketamine | Total
Number analyzed (Participants) | 9 | 16 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 16 | 25
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 16 | 25
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 8 | 11 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 16 | 25

OUTCOME MEASURES:

1. Primary Outcome: TcCO2 Above 50
Description: % Time Tosca Monitor (TcCO2) above 50. A TcCo2 above 50 is indicative of hypoventilation.
Time Frame: Intraoperative, an average of about 1 and 1/2 hours.
Measure: Mean (Standard Deviation); unit: Percent time intraoperatrive
Arm/Group | Ketamine Group | No Ketamine
Number analyzed (Participants) | 8 | 15
Percent time intraoperatrive | 39 (26.54) | 30.8 (26.14)

ADVERSE EVENTS:
Time Frame: 24 hours
Groups:
- No Ketamine Added to Anesthesia Regimen: No ketamine added to the patients anesthesia regimen
- Ketamine Group: Ketamine group: Ketamine group: ketamine bolus of 0.25mg/kg followed by an infusion set at 1.5 mcg /kg/min.
Arm/Group | No Ketamine Added to Anesthesia Regimen | Ketamine Group
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/9
Other Adverse Events (participants affected / at risk) | 0/16 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No